CLINICAL TRIAL: NCT06746454
Title: Gender-Specific Effects of Different Focus of Attention Instructions on Landing Technique, Alignment, and Joint Position Sense in Semi-Professional Volleyball Players
Brief Title: The Gender-Specific Effect of Different Instruction Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Pelin Pişirici, Assistant Professor, PT, PhD, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: OS-GenderF
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Sports Injury
Keywords: motor learning; proprioception; volleyball; knee valgus; drop vertical jump test
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Intervention Model Description: Randomized, single-blind, prospective study
Who Masked: Outcomes Assessor
Masking Description: Randomization was gender specific. Female participants were randomized to the verbal training group with combined attentional focus instruction (VFIT) and the visual training group with video instruction (VGE) by asking them to draw a paper from a black bag filled with papers with the names of both groups. For male participants, randomization was performed with a different black bag with the same characteristics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video Instructed Training Group (Experimental): Video Instructed Training Group Before the study is conducted, the expert video that will be used for the VI group instructions will be created. The expert video was created with an athlete with a LESS score of less than 4 and an FPPA of less than 10 who performs a DVJ task following the instructions. The video recording was used only for the video group instructions.
  Interventions: Other: Video Instructed Training Group
- Verbal Combined Focus Instructed Training Group (Experimental): Participants will be given combined verbal instruction such as "Focus on how hard you push yourself off the ground after the jump and how quickly you straighten your knees during this push", in which internal and external focus directions were given simultaneously.
  Interventions: Other: Verbal Combined Focus Instructed Training Group

INTERVENTIONS:
Other: Video Instructed Training Group — "Pre-test" measurements were taken to determine the baseline values of the athletes before the training packages specific to their group. The pre-test measurements included a landing error scoring system, knee position error sense, and frontal plane projection angle. After the pre-test measurements, 2 training packages with special instructions were performed for the video instructed training (VIT) group. The special instruction for the VIT group included a previously prepared video of a successful vertical jump landing task. This video was shown to the VIT group. Immediately after the training packages, post-test measurements were taken. The post-test measurements included the same tests as the pre-test measurements. A follow-up test was taken 7 days after the measurements. The follow-up test included the same measurements as in the pre-test and post-test phases.
  Arms: Video Instructed Training Group
Other: Verbal Combined Focus Instructed Training Group — "Pre-test" measurements were taken to determine the baseline values of the athletes before the training packages specific to their group. The pre-test measurements included landing error scoring system, knee position error sense, and frontal plane projection angle. After the pretest measurements, 2 training packages with specific instructions were performed for the CSE group. The special instruction given to the CSE group consisted of the following sentence, which included the both internal and external focus of attention; "focus on how hard you push yourself off the ground and how fast you straighten your knees during this push-off". Immediately after the training packages, post-test measurements were taken. The post-test measurements included the same tests as the pre-test measurements. A follow-up test was taken 7 days after the measurements. The follow-up test included the same measurements as in the pre-test and post-test phases.
  Arms: Verbal Combined Focus Instructed Training Group

SUMMARY:
Feedback is incorporated into training programs to prevent injuries. The superiority of several feedback techniques is still debated and there is a need for gender specific studies. The main aim of the study was to investigate the gender-specific effectiveness of two different feedback techniques (combined verbal training with internal and external focus feedback and video training with instructional feedback) on the landing technique after vertical jump, frontal plane projection angle, and joint position sense in male and female volleyball players with asymptomatic knee valgus. In addition, the continuity of potential positive results in a retention test performed one week after the test session will be evaluated.

DETAILED DESCRIPTION:
Prevention of knee injuries in sports, especially in contact sports, is important for both the health of the athlete and the success of the team. Volleyball injuries are seen in the knee region with a rate of 23.66%. Jumping to the ground is a common injury mechanism in both genders.

The anatomical and physiological differences of young athletes make them more prone to these injuries. Anatomical variations, hormonal effects, and neuromuscular control problems are among the factors that increase the likelihood of these injuries.

Male athletes are considered to be prone to ACL injuries due to hormonal changes that occur during puberty. Furthermore, it has been reported that men are more frequently exposed to ankle and knee injuries in sports such as volleyball.

In terms of female athletes, it has been observed that hormonal fluctuations may increase the risk of injury by affecting the structure and durability of connective tissue. It has been stated that changes in various hormones during the menstrual cycle cause ligaments to become looser. This is a factor that increases the risk of injury during physical activities.

Current rehabilitation programs focus on neuromuscular training programs to prevent negative movement patterns and increase proper movement control. Neuromuscular training programs are exercise approaches that aim to improve skills such as motor control, strength, balance, coordination, and proprioception. These programs strengthen balance and stability, especially in the lower extremities, allowing athletes to perform movements such as sudden changes of direction, jumping, and landing more safely.

However, there is a need to increase the effectiveness of these neuromuscular training programs to have a more significant impact on ACL injury rates. Therefore, the use of motor learning strategies and neuromuscular training programs with adequate and correct techniques in the rehabilitation of athletes still needs to be investigated.

The incorporation of feedback instructions into injury programs is frequently reported in the current literature, and the common denominator that studies have found is the use of clear directives and specific instructions regarding the desired landing position.

Motor skills can be learned with an internal focus of attention or with an external focus of attention. Although the difference between these instructions may seem insignificant, externally focused training has resulted in better performance, retention, transfer and greater movement automaticity. Furthermore, other studies have shown that internal focus of attention instructions are superior to external focus of attention in motor learning in various disciplines. Recent literature highlights the necessity of using both feedback techniques at the same time as combined.

Observation is an effective method to improve motor skill learning. Observing the data given with video feedback and imitating it by copying the body movements. The usage of video feedback is beneficial by contributing to lower limb dynamics during landing movements after jumping. Further studies are needed to examine the effect of video feedback on different genders.

The main aim of the study was to investigate the gender-specific effectiveness of two different feedback techniques (combined verbal training with internal and external focus feedback and video training with instructional feedback) on the landing technique after the vertical jump, frontal plane projection angle, and joint position sense in male and female volleyball players with asymptomatic knee valgus.

However, there is a need to increase the effectiveness of these neuromuscular training programs to have a more significant impact on ACL injury rates. Therefore, the use of motor learning strategies and neuromuscular training programs with adequate and correct techniques in the rehabilitation of athletes still needs to be investigated.

The incorporation of feedback instructions into injury programs is frequently reported in the current literature, and the common denominator that studies have found is the use of clear directives and specific instructions regarding the desired landing position.

Motor skills can be learned with an internal focus of attention or with an external focus of attention. Although the difference between these instructions may seem insignificant, externally focused training has been shown to result in better performance, retention, transfer, and greater movement automaticity. Furthermore, other studies have shown that the internal focus of attention instructions is superior to the external focus of attention in motor learning in various disciplines. Recent literature highlights the necessity of using both feedback techniques at the same time as combined.

Observation is an effective method to improve motor skill learning. Observing the data given with video feedback and imitating it by copying the body movements. The usage of video feedback is beneficial by contributing to lower limb dynamics during landing movements after jumping. Further studies are needed to examine the effect of video feedback on different genders.

The main aim of the study was to investigate the gender-specific effectiveness of two different feedback techniques (combined verbal training with internal and external focus feedback and video training with instructional feedback) on the landing technique after the vertical jump, frontal plane projection angle, and joint position sense in male and female volleyball players with asymptomatic knee valgus.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-24
* Becoming a minor volleyball player
* Volunteers must not have suffered any trunk or lower extremity injuries in the last 6 months before participation in the study.
* Having a frontal plane projection angle greater than 10° during the single-leg squat test

Exclusion Criteria:

* Having experienced a trunk or lower extremity injury in the last 6 months before the date of study
* Having a history of fracture or dislocation in the lower extremity
* Having suffered from back pain in the past years
* Having a musculoskeletal system abnormality
* Being unable to perform functional tasks (visual, auditory, vestibular or neurological impairment)
* Being pregnant
* Having malignancy and metabolic diseases

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2024-11-05 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Landing Error Scoring System (LESS) Measurement | baseline, immediately after the intervention, one week after the baseline
  Two standard video cameras capture the frontal plane and sagittal plane view of each subject as they perform the test procedures (jumping from 30 cm height box). The participant's LESS score represents excellent (LESS score <4), good (LESS score >4 to 5), fair (LESS score >5 to 6) and poor (LESS score >6) jumping technique.

SECONDARY OUTCOMES:
Frontal Plan Projection Angle (FPPA) Measurement | baseline, immediately after the intervention, one week after the baseline
  During the frontal plane projection angle (FPPA) measurement, a straight line will be drawn from the anterior superior spina iliaca along the femur to the midpoint of the patella, and the midpoint of the ankle will be determined as the reference point by a straight line drawn from the midpoint of the patella. Participants will stand with their feet aligned in the sagittal plane and their arms crossed across their chests. By prior instruction, subjects will be asked to squat up to 60º knee flexion in a controlled manner without losing their balance, before returning to the starting position. Digital recordings of the frontal plane will be made while individuals perform a single-leg squat test at 60º knee flexion 3 times. The FPPA degree is measured from the medial aspect of the knee and calculated by subtracting 360. FPPA of 195° and above will be considered pathological.
Knee Joint Position Sense (KJPS) Measurement | baseline, immediately after the intervention, one week after the baseline
  Participants are initially placed in a sitting position in 90° knee flexion. Participants' eyes are covered with a mask to block visual input. The smartphone that will perform the measurement is fixed to the participants' lower limb (15 cm from the apex of the fibular head) with a Velcro strap. From the starting position (90 knee flexion), the participants' knee is placed by the researcher at a target joint angle of 45. Participants actively hold the knee at the 45 target joint angle for five seconds to understand the exact angle of the knee. After these five seconds, the participants actively return their knee to the starting position and the researcher shows the target angle to the participant three times. With the command given by the researcher, the participants are directed to extend their knees as close as possible to the target joint angle without any external stimulation or assistance. Participants perform 3 trials and try to maintain the estimated position for 3 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Oktay Şenozan, PT, Principal Investigator — Bahcesehir University, Graduate Education Institute, Physiotherapy and Rehabilitation, Master of Science Program; Pelin Pişirici, PT, PhD, Study Director — Bahcesehir University, Faculty of Health Sciences
Locations (1):
- Smyrna Sports Club, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No